CLINICAL TRIAL: NCT02164513
Title: A Phase III, 52 Week, Randomized, Double-blind, 3-arm Parallel Group Study, Comparing the Efficacy, Safety and Tolerability of the Fixed Dose Triple Combination FF/UMEC/VI With the Fixed Dose Dual Combinations of FF/VI and UMEC/VI, All Administered Once-daily in the Morning Via a Dry Powder Inhaler in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A Study Comparing the Efficacy, Safety and Tolerability of Fixed Dose Combination (FDC) of FF/UMEC/VI With the FDC of FF/VI and UMEC/VI; Administered Once-daily Via a Dry Powder Inhaler (DPI) in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116855
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; umeclidinium; fluticasone furoate; vilanterol; triple therapy; exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fluticasone furoate/umeclidinium bromide/vilanterol (Experimental): Eligible Subjects completing 2-weeks run-in period will receive FF/UMEC/VI 100 mcg/62.5 mcg/25 mcg QD (morning) for a period of 52 weeks via DPI
  Interventions: Drug: fluticasone furoate (FF); Drug: vilanterol (VI); Drug: umeclidinium bromide (UMEC)
- fluticasone furoate/vilanterol (Experimental): Eligible Subjects completing 2-weeks run-in period will receive FF/VI 100 mcg/25 mcg QD (morning) for a treatment period of 52 weeks via DPI)
  Interventions: Drug: fluticasone furoate (FF); Drug: vilanterol (VI)
- umeclidinium bromide/vilanterol (Experimental): Eligible Subjects completing 2-weeks run-in period will receive UMEC/VI 62.5 mcg/25 mcg QD (morning) for a treatment period of 52 weeks via DPI
  Interventions: Drug: vilanterol (VI); Drug: umeclidinium bromide (UMEC)

INTERVENTIONS:
Drug: fluticasone furoate (FF) — FF will be available in combination as dry powder for inhalation as FF/UMEC/VI 100 mcg/62.5 mcg/25 mcg and FF/VI 100 mcg/25 mcg
  Arms: fluticasone furoate/umeclidinium bromide/vilanterol; fluticasone furoate/vilanterol
Drug: vilanterol (VI) — VI will be available in combination as dry powder for inhalation as FF/UMEC/VI 100 mcg/62.5 mcg/25 mcg, FF/VI 100 mcg/25 mcg and UMEC/VI 62.5 mcg/25 mcg
Drug: umeclidinium bromide (UMEC) — UMEC will be available in combination as dry powder for inhalation as FF/UMEC/VI 100 mcg/62.5 mcg/25 mcg, and UMEC/VI 62.5 mcg/25 mcg
  Arms: fluticasone furoate/umeclidinium bromide/vilanterol; umeclidinium bromide/vilanterol

SUMMARY:
The study evaluates the efficacy of fluticasone furoate/umeclidinium bromide/vilanterol (FF/UMEC/VI) to reduce the annual rate of moderate and severe exacerbations compared with dual therapy of FF/VI or UMEC/VI in subjects with COPD. Published studies which assessed the use of an 'open' triple therapy (use of Inhaled Corticosteroid [ICS]/ Long-acting Muscarinic Receptor Antagonists [LAMA])/ Long Acting Beta-Agonist [LABA] delivered via multiple inhalers) in moderate-severe COPD patients, reported improvements in lung function, Health Related Quality of Life (HRQoL), hospitalization rates and rescue medication use, compared to dual therapy (ICS/LABA) or LAMA alone. These studies have also shown similar safety profile with dual or monotherapy doses for periods of up to one year. Given the clinical experience with FF, UMEC and VI, and that the associated risks with these compounds are anticipated from their known pharmacology, the potential benefit of a new therapy option in patients with moderate to severe COPD supports the further development of the closed triple combination (delivered via one inhaler). In the current study subjects meeting all inclusion/exclusion criteria will complete 2-week run-in period; 52 week treatment period and a 1-week safety follow-up period. Eligible subjects will be randomized to one of the following double-blind treatment groups FF/UMEC/VI 100 micrograms (mcg)/62.5 mcg/25 mcg once daily (QD), FF/VI 100 mcg/25 mcg QD, or UMEC/VI 62.5 mcg/25 mcg QD

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: A signed and dated written informed consent prior to study participation
* Type of subject: Outpatient
* Age: Subjects 40 years of age or older at Visit 1
* Gender: Male or female subjects. A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g. age appropriate, > 45 years, in the absence of hormone replacement therapy OR Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e. in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to safety follow-up contact): Abstinence; Oral Contraceptive, either combined or progestogen alone; Injectable progestogen; Implants of levonorgestrel; Estrogenic vaginal ring; Percutaneous contraceptive patches; Intrauterine device (IUD) or intrauterine system (IUS); Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records. Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* COPD Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years at screening (visit 1) [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Note: Pipe and/or cigar use cannot be used to calculate pack-year history
* Severity of COPD symptoms: A score of >=10 on the COPD Assessment Test (CAT) at screening
* Severity of COPD Disease: A post-albuterol/salbutamol FEV1/ Forced Vital Capacity (FVC) ratio of <0.70 at Screening
* Existing COPD maintenance treatment: Subject must be receiving daily maintenance treatment for their COPD for at least 3 months prior to Screening. Note: Subjects receiving only Pro re nata (PRN) COPD medications are not eligible
* History of Exacerbations: Subjects must demonstrate: a post-bronchodilator FEV1 <50% predicted normal and a documented history of >= 1 moderate or severe COPD exacerbation in the previous 12 months OR a post-bronchodilator 50% <=FEV1 < 80% predicted normal and a documented history of >= 2 moderate exacerbations or a documented history of >=1 severe COPD exacerbation (hospitalized) in the previous 12 months. Note: Percent predicted will be calculated using the European Respiratory Society Global Lung Function Initiative reference equations. Note: A documented history of a COPD exacerbation (e.g., medical record verification) is a medical record of worsening COPD symptoms that required systemic/oral corticosteroids and/or antibiotics (for a moderate exacerbation) or hospitalization (for a severe exacerbation). Prior use of antibiotics alone does not qualify as an exacerbation history unless the use was associated with treatment of worsening symptoms of COPD, such as increased dyspnea, sputum volume, or sputum purulence (color). Subject verbal reports are not acceptable
* Liver function tests: alanine aminotransferase (ALT) <2x upper limit of normal (ULN); alkaline phosphatase <=1.5xULN; bilirubin <=1.5xULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study
* Asthma: Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD)
* Alpha1-antitrypsin deficiency: Subjects with Alpha1-antitrypsin deficiency as the underlying cause of COPD
* Other respiratory disorders: Subjects with active tuberculosis, lung cancer, significant bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases
* Lung resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening
* Risk Factors for Pneumonia: immune suppression (e.g. human immunodeficiency virus [HIV], Lupus) or other risk factors for pneumonia (e.g. neurological disorders affecting control of the upper airway, such as Parkinson's Disease, Myasthenia Gravis). Patients at potentially high risk (e.g. very low BMI, severely malnourished, or very low FEV1) will only be included at the discretion of the Investigator
* Pneumonia and/or moderate or severe COPD exacerbation that has not resolved at least 14 days prior to Screening and at least 30 days following the last dose of oral/systemic corticosteroids (if applicable). In addition, any subject that experiences pneumonia and/or moderate or severe COPD exacerbation during the run-in period will be excluded
* Other Respiratory tract infections that have not resolved at least 7 days prior to screening
* Abnormal Chest x-ray(CXR): Chest x-ray (posteroanterior and lateral) reveals evidence of pneumonia or a clinically significant abnormality not believed to be due to the presence of COPD, or another condition that would hinder the ability to detect an infiltrate on CXR (e.g. significant cardiomegaly, pleural effusion or scarring). All subjects will have a chest x-ray at Screening Visit 1 (or historical radiograph or computerised tomography (CT) scan obtained within 3 months prior to screening) that will be over-read by a central vendor. Note: Subjects who have experienced pneumonia and/or moderate or severe COPD exacerbation within 3 months of screening must provide a post pneumonia/exacerbation chest x-ray to be over-read by the central vendor or have a chest x-ray conducted at screening. For sites in Germany: If a chest x-ray (or CT scan) within 3 months prior to Screening (Visit 1) is not available, approval to conduct a diagnostic chest x-ray will need to be obtained from the Federal Office for Radiation Protection (Bundesamt für Strahlenschutz [BfS])
* Other diseases/abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study
* Unstable liver disease as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice, cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Note: Chronic stable hepatitis B and C are acceptable if the subject otherwise meets entry criteria
* Unstable or life threatening cardiac disease: subjects with any of the following at Screening (Visit 1) would be excluded: Myocardial infarction or unstable angina in the last 6 months; Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months; New York Heart Association (NYHA) Class IV Heart failure
* Abnormal and clinically significant 12-Lead Electrocardiogram (ECG) finding: Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. The Principal Investigator will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. An abnormal and clinically significant finding that would preclude a subject from entering the trial is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following: atrial fibrillation (AF) with rapid ventricular rate >120 beats per minute); sustained or nonsustained ventricular tachycardia (VT); Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted); QT interval corrected for heart rate (QTcF) >=500 milliseconds (msec) in patients with QRS <120 msec and QTcF >=530 msec in patients with QRS >=120 msec
* Contraindications: A history of allergy or hypersensitivity to any corticosteroid, anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the Investigator contraindicates study participation
* Cancer: Subjects with carcinoma that has not been in complete remission for at least 5 years. Subjects who have had carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded based on the 5 year waiting period if the subject has been considered cured by treatment
* Oxygen therapy: Use of long-term oxygen therapy (LTOT) described as resting oxygen therapy >3 Liter/minute (L/min) (Oxygen use =<3L/min flow is not exclusionary)
* Medication prior to spirometry: Subjects who are medically unable to withhold their albuterol/salbutamol for the 4-hour period required prior to spirometry testing at each study visit
* Pulmonary rehabilitation: Subjects who have participated in the acute phase of a Pulmonary Rehabilitation Program within 4 weeks prior to Screening or subjects who plan to enter the acute phase of a Pulmonary Rehabilitation Program during the study. Subjects who are in the maintenance phase of a Pulmonary Rehabilitation Program are not excluded
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years
* Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study
* Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study
* Inability to read: In the opinion of the Investigator, any subject who is unable to read and/or would not be able to complete study related materials
* Medication prior to screening: Use of the following medications within the following time intervals prior to Screening (Visit 1) or during the study: Long term antibiotic therapy Subjects receiving antibiotics for long term therapy are not eligible for the study (Antibiotics are allowed for the short term treatment of an exacerbation or for short term treatment of other acute infections during the study); Systemic, Oral, parenteral corticosteroids 30 days (Except during the study oral/systemic corticosteroids may be used to treat COPD exacerbations/pneumonia) Intra-articular injections are allowed; Any other investigational drug (30 days or 5 half lives whichever is longer)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10355 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (737):
- United States (229):
  - GSK Investigational Site, Athens, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Florence, Alabama
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Muscle Shoals, Alabama
  - GSK Investigational Site, Sheffield, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Flagstaff, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Arcadia, California
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Escondido, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Mission Hills, California
  - GSK Investigational Site, Modesto, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, Reseda, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Danbury, Connecticut
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, West Haven, Connecticut
  - GSK Investigational Site, Bay Pines, Florida
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Celebration, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Edgewater, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Leesburg, Florida
  - GSK Investigational Site, Loxahatchee Groves, Florida
  - GSK Investigational Site, Maitland, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Oviedo, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Ponte Vedra Beach, Florida
  - GSK Investigational Site, Port Charlotte, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Adairsville, Georgia
  - GSK Investigational Site, Athens, Georgia
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Conyers, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Duluth, Georgia
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Rincon, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Elk Grove Village, Illinois
  - GSK Investigational Site, Gillespie, Illinois
  - GSK Investigational Site, Hines, Illinois
  - GSK Investigational Site, O'Fallon, Illinois
  - GSK Investigational Site, Oak Park, Illinois
  - GSK Investigational Site, Quincy, Illinois
  - GSK Investigational Site, Winfield, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Franklin, Indiana
  - GSK Investigational Site, Greenfield, Indiana
  - GSK Investigational Site, Muncie, Indiana
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Olathe, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Fort Mitchell, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Crowley, Louisiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Hollywood, Maryland
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Pittsfield, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Duluth, Minnesota
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, Fridley, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Woodbury, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Fremont, Nebraska
  - GSK Investigational Site, Grand Island, Nebraska
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Reno, Nevada
  - GSK Investigational Site, Marlton, New Jersey
  - GSK Investigational Site, Moorestown, New Jersey
  - GSK Investigational Site, Neptune City, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Bronxville, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Calabash, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Hendersonville, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Lexington, North Carolina
  - GSK Investigational Site, Mooresville, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Whiteville, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Marion, Ohio
  - GSK Investigational Site, Middleburg Heights, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Wooster, Ohio
  - GSK Investigational Site, Corvallis, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Downingtown, Pennsylvania
  - GSK Investigational Site, Doylestown, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Johnstown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Phoenixville, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Tipton, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Fort Mill, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Hendersonville, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Edinburg, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Gonzales, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Kerrville, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sealy, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Renton, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane Valley, Washington
  - GSK Investigational Site, Tacoma, Washington
- Argentina (27):
  - GSK Investigational Site, Bahía Blanca, Buenos Aires
  - GSK Investigational Site, CABA, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Florida, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Nueve de Julio, Buenos Aires
  - GSK Investigational Site, Paraná, Buenos Aires
  - GSK Investigational Site, Vicente López, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Concepción del Uruguay, Entre Ríos Province
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Berazategui
  - GSK Investigational Site, Berazategui, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Ciudad Autonoma de Buenis Aires
  - GSK Investigational Site, Coronel Suárez
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Monte Grande
  - GSK Investigational Site, Salta
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, Santa Fe
  - GSK Investigational Site, Santa Rosa
- Australia (16):
  - GSK Investigational Site, Concord, New South Wales
  - GSK Investigational Site, Gosford, New South Wales
  - GSK Investigational Site, Maroubra, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Cairns, Queensland
  - GSK Investigational Site, Carina Heights, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Daw Park, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Footscray, Victoria
  - GSK Investigational Site, Frankston, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Hamilton, Victoria
  - GSK Investigational Site, Murdoch, Western Australia
  - GSK Investigational Site, Nedlands, Western Australia
  - GSK Investigational Site, Liverpool
- Austria (5):
  - GSK Investigational Site, Feldbach
  - GSK Investigational Site, Feldkirch
  - GSK Investigational Site, Grieskirchen
  - GSK Investigational Site, Thalheim bei Wels
  - GSK Investigational Site, Vienna
- Belgium (15):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Erpent
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Gilly
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Malmedy
  - GSK Investigational Site, Mechelen
  - GSK Investigational Site, Montigny-le-Tilleul
  - GSK Investigational Site, Ostend
  - GSK Investigational Site, Roeselaere
  - GSK Investigational Site, Turnhout
- Brazil (6):
  - GSK Investigational Site, Recife, Pernambuco
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Blumenau, Santa Catarina
  - GSK Investigational Site, Florianópolis, Santa Catarina
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Canada (18):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Sherwood Park, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Cornwall, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Chile (10):
  - GSK Investigational Site, Curicó, Maule Region
  - GSK Investigational Site, Talca, Maule Region
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Concepción, Región Del Biobio
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Talcahuano
  - GSK Investigational Site, Viña del Mar
- China (25):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Zhanjiang, Guangdong
  - GSK Investigational Site, Nanning, Guangxi
  - GSK Investigational Site, Haikou, Hainan
  - GSK Investigational Site, Shijiazhuang, Hebei
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Nanchang, Jiangxi
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Yinchuan, Ningxia
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Qingdao, Shandong
  - GSK Investigational Site, Taiyuan, Shanxi
  - GSK Investigational Site, Xian, Shanxi
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Fuzhou
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Wuxi
- Colombia (3):
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Medellín
- Czechia (13):
  - GSK Investigational Site, Benešov
  - GSK Investigational Site, Brandýs nad Labem
  - GSK Investigational Site, Cvikov
  - GSK Investigational Site, Holešov
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Jaroměř
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Tábor
  - GSK Investigational Site, Teplice
  - GSK Investigational Site, Třebíč
- Denmark (8):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Aarhus C
  - GSK Investigational Site, Hellerup
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Kolding
  - GSK Investigational Site, Odense C
  - GSK Investigational Site, Roskilde
  - GSK Investigational Site, Sønderborg
- Finland (6):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jyväskylä
  - GSK Investigational Site, Lohja
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (19):
  - GSK Investigational Site, Bayonne
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Briis-sous-Forge
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Le Mans
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montauban
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Perpignan
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Pringy
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (83):
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Leonberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Wiesloch, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Bad Woerrishofen, Bavaria
  - GSK Investigational Site, Bamberg, Bavaria
  - GSK Investigational Site, Dachau, Bavaria
  - GSK Investigational Site, Dillingen an der Donau, Bavaria
  - GSK Investigational Site, Donaustauf, Bavaria
  - GSK Investigational Site, Garmisch-Partenirchen, Bavaria
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Landsberg am Lech, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Neu-Ulm, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Rosenheim, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Rathenow, Brandenburg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Bensheim, Hesse
  - GSK Investigational Site, Frankenberg, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Fuldatal, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Offenbach, Hesse
  - GSK Investigational Site, Rodgau, Hesse
  - GSK Investigational Site, Rüsselsheim am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Peine, Lower Saxony
  - GSK Investigational Site, Wardenburg, Lower Saxony
  - GSK Investigational Site, Bad Lippspringe, North Rhine-Westphalia
  - GSK Investigational Site, Bergisch Gladbach, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Düren, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Freudenberg, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Gummersbach, North Rhine-Westphalia
  - GSK Investigational Site, Hagen, North Rhine-Westphalia
  - GSK Investigational Site, Kleve, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Ratingen, North Rhine-Westphalia
  - GSK Investigational Site, Rheine, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Warendorf, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Bernkastel-Kues, Rhineland-Palatinate
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Neuwied, Rhineland-Palatinate
  - GSK Investigational Site, Wissen, Rhineland-Palatinate
  - GSK Investigational Site, Saarbrücken, Saarland
  - GSK Investigational Site, Auerbach, Saxony
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halberstadt, Saxony-Anhalt
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Hettstedt, Saxony-Anhalt
  - GSK Investigational Site, Teuchern, Saxony-Anhalt
  - GSK Investigational Site, Zerbst, Saxony-Anhalt
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Reinfeld, Schleswig-Holstein
  - GSK Investigational Site, Schleswig, Schleswig-Holstein
  - GSK Investigational Site, Gera, Thuringia
  - GSK Investigational Site, Saalfeld, Thuringia
  - GSK Investigational Site, Schmölln, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Deggendorf
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Witten
- Hong Kong (5):
  - GSK Investigational Site, Kwun Tong
  - GSK Investigational Site, Lai Chi Kok
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
  - GSK Investigational Site, Tuenmen
- Israel (11):
  - GSK Investigational Site, Afula
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
  - GSK Investigational Site, Zrifin
- Japan (33):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Toyama
  - GSK Investigational Site, Wakayama
  - GSK Investigational Site, Yamagata
  - GSK Investigational Site, Yamanashi
- Netherlands (23):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Assen
  - GSK Investigational Site, Beek
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Dordrecht
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Helmond
  - GSK Investigational Site, Hoofddorp
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Kloosterhaar
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Sneek
  - GSK Investigational Site, Spijkenisse
  - GSK Investigational Site, Veldhoven
  - GSK Investigational Site, Zutphen
  - GSK Investigational Site, Zwolle
- New Zealand (5):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Newtown, Wellington
  - GSK Investigational Site, Tauranga
  - GSK Investigational Site, Wellington
- Norway (8):
  - GSK Investigational Site, Bodø
  - GSK Investigational Site, Fredrikstad
  - GSK Investigational Site, Hakadal
  - GSK Investigational Site, Kløfta
  - GSK Investigational Site, Levanger
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Trondheim
- Peru (4):
  - GSK Investigational Site, Pueblo Libre, Lima region
  - GSK Investigational Site, San Martín de Porres, Lima region
  - GSK Investigational Site, San Miguel, Lima region
  - GSK Investigational Site, Lima
- Philippines (5):
  - GSK Investigational Site, Caloocan
  - GSK Investigational Site, Iloilo City
  - GSK Investigational Site, Jaro, Iloilo City
  - GSK Investigational Site, Pasig
  - GSK Investigational Site, Quezon City
- Poland (6):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Zgierz
- Puerto Rico (4):
  - GSK Investigational Site, Guaynabo
  - GSK Investigational Site, Mayagüez
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, San Juan
- Romania (7):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Brăila
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Comuna Alexandru Cel Bun
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Râmnicu Vâlcea
- Russia (27):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Belgorod
  - GSK Investigational Site, Blagoveshchensk
  - GSK Investigational Site, Chita
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Petrozavodsk
  - GSK Investigational Site, Pyatigorsk
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ulan-Ude
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Veliky Novgorod
  - GSK Investigational Site, Vladimir
  - GSK Investigational Site, Vladivostok
  - GSK Investigational Site, Volgodonsk
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Vsevolozhsk, Leningrad Region
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- GSK Investigational Site, Singapore, Singapore
- South Africa (19):
  - GSK Investigational Site, Benoni, Gauteng
  - GSK Investigational Site, Boksburg, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Val de Grace, Pretoria, Gauteng
  - GSK Investigational Site, Middelburg, Mpumalanga
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Boksburg North
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, CapeTown
  - GSK Investigational Site, Durban
  - GSK Investigational Site, eManzimtoti
  - GSK Investigational Site, Gatesville
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Korsten
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Paarl
  - GSK Investigational Site, Panorama
  - GSK Investigational Site, Tygerberg
- South Korea (8):
  - GSK Investigational Site, Bucheon City, Gyenggi-do
  - GSK Investigational Site, Cheongju-si, Chungcheongbuk-do
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
- Spain (43):
  - GSK Investigational Site, Marbella - Málaga, Andalusia
  - GSK Investigational Site, Laredo, Cantabria
  - GSK Investigational Site, Torrelavega, Cantabria
  - GSK Investigational Site, Badalona, Catalonia
  - GSK Investigational Site, (Badalona) Barcelona
  - GSK Investigational Site, (Barakaldo) Vizcaya
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Alzira/Valencia
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Basurto/Bilbao
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Centelles (Barcelona)
  - GSK Investigational Site, Coslada
  - GSK Investigational Site, Girona
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Mérida (Badajoz)
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Peralada( Girona)
  - GSK Investigational Site, Petrer/Alicante
  - GSK Investigational Site, Ponferrada (León)
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Sagunto/Valencia
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, San Sebastián de los Reyes
  - GSK Investigational Site, Sant Joan d'Alacant
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Tarragona
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Vizcaya
  - GSK Investigational Site, Zaragoza
- Sweden (9):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Höllviken
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Luleå
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Östersund
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- Thailand (7):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Muang
  - GSK Investigational Site, Nakhon Ratchasima
  - GSK Investigational Site, Nan
  - GSK Investigational Site, Songkhla
- Turkey (Türkiye) (4):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Izmir
  - GSK Investigational Site, Mersin
- Ukraine (7):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Mykolayiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Sumy
  - GSK Investigational Site, Vinnytsia
- United Kingdom (16):
  - GSK Investigational Site, Exeter, Devon
  - GSK Investigational Site, Wishaw, Lanarkshire
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, High Heaton, Newcastle Upon Tyne, Tyne & Wear
  - GSK Investigational Site, Bradford-on-Avon, Wiltshire
  - GSK Investigational Site, Baillieston, Glasgow
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Chester
  - GSK Investigational Site, Crawley
  - GSK Investigational Site, Crownhill, Plymouth
  - GSK Investigational Site, Dundee, Scotland
  - GSK Investigational Site, Sidcup, Kent
  - GSK Investigational Site, Stockton-on-Tees
  - GSK Investigational Site, Trowbridge
- Vietnam (2):
  - GSK Investigational Site, Hà Nội
  - GSK Investigational Site, Ho Chi Minh City

REFERENCES:
- [Derived] Risebrough NA, Mursleen S, Ndirangu K, Shah D, Martin A, Schroeder M, Ismaila AS. The long-term clinical and economic benefits of treating advanced COPD patients with single-inhaler triple therapy in Quebec, Canada - The IMPACT trial. Respir Med. 2024 Sep;231:107694. doi: 10.1016/j.rmed.2024.107694. Epub 2024 Jun 4. PMID 38844004
- [Derived] Aggarwal B, Jones P, Casas A, Gomes M, Juthong S, Litewka D, Ong-Dela Cruz B, Ramirez-Venegas A, Sayiner A, van Hasselt J, Compton C, Tombs L, Weng S, Levy G. Association between Increased Risk of Pneumonia with ICS in COPD: A Continuous Variable Analysis of Patient Factors from the IMPACT Study. Pulm Ther. 2024 Jun;10(2):183-192. doi: 10.1007/s41030-024-00255-1. Epub 2024 Mar 6. PMID 38446336
- [Derived] Verstraete K, Gyselinck I, Huts H, Das N, Topalovic M, De Vos M, Janssens W. Estimating individual treatment effects on COPD exacerbations by causal machine learning on randomised controlled trials. Thorax. 2023 Oct;78(10):983-989. doi: 10.1136/thorax-2022-219382. Epub 2023 Apr 3. PMID 37012070
- [Derived] Bardsley S, Criner GJ, Halpin DMG, Han MK, Hanania NA, Hill D, Lange P, Lipson DA, Martinez FJ, Midwinter D, Siler TM, Singh D, Wise RA, van Zyl-Smit RN, Berkman N. Single-inhaler triple therapy fluticasone furoate/umeclidinium/vilanterol versus dual therapy in current and former smokers with COPD: IMPACT trial post hoc analysis. Respir Med. 2022 Dec;205:107040. doi: 10.1016/j.rmed.2022.107040. Epub 2022 Nov 11. PMID 36470149
- [Derived] Dransfield MT, Criner GJ, Halpin DMG, Han MK, Hartley B, Kalhan R, Lange P, Lipson DA, Martinez FJ, Midwinter D, Singh D, Wise R, Kunisaki KM. Time-Dependent Risk of Cardiovascular Events Following an Exacerbation in Patients With Chronic Obstructive Pulmonary Disease: Post Hoc Analysis From the IMPACT Trial. J Am Heart Assoc. 2022 Sep 20;11(18):e024350. doi: 10.1161/JAHA.121.024350. Epub 2022 Sep 14. PMID 36102236
- [Derived] Thompson PJ, Criner GJ, Dransfield MT, Halpin DMG, Han MK, Lipson DA, Maghzal GJ, Martinez FJ, Midwinter D, Singh D, Tombs L, Wise RA. Effect of chronic mucus hypersecretion on treatment responses to inhaled therapies in patients with chronic obstructive pulmonary disease: Post hoc analysis of the IMPACT trial. Respirology. 2022 Dec;27(12):1034-1044. doi: 10.1111/resp.14339. Epub 2022 Aug 15. PMID 35970518
- [Derived] Thomashow B, Stiegler M, Criner GJ, Dransfield MT, Halpin DMG, Han MK, Lange P, Martinez FJ, Midwinter D, Singh D, Tabberer M, Wise RA, Lipson DA, Jones P. Higher COPD Assessment Test Score Associated With Greater Exacerbations Risk: A Post Hoc Analysis of the IMPACT Trial. Chronic Obstr Pulm Dis. 2022 Jan 27;9(1):68-79. doi: 10.15326/jcopdf.2021.0259. PMID 34972260
- [Derived] Bafadhel M, Barnes N, Bourke SC, Compton C, Criner GJ, Dransfield MT, Halpin DMG, Han MK, Hartley B, Jones CE, Lange P, Lettis S, Lipson DA, Lomas DA, Martin N, Martinez FJ, Wise R, Singh D. A single blood eosinophil count measurement is as good as two for prediction of ICS treatment response in the IMPACT trial. Eur Respir J. 2021 Sep 23;58(3):2004522. doi: 10.1183/13993003.04522-2020. Print 2021 Sep. No abstract available. PMID 34385263
- [Derived] Singh D, Criner GJ, Dransfield MT, Halpin DMG, Han MK, Lange P, Lettis S, Lipson DA, Mannino D, Martin N, Martinez FJ, Miller BE, Wise R, Zhu CQ, Lomas D. InforMing the PAthway of COPD Treatment (IMPACT) trial: fibrinogen levels predict risk of moderate or severe exacerbations. Respir Res. 2021 Apr 28;22(1):130. doi: 10.1186/s12931-021-01706-y. PMID 33910578
- [Derived] Halpin DMG, Criner GJ, Dransfield MT, Han MK, Hartley B, Harvey C, Jones CE, Kato M, Lange P, Lettis S, Lomas DA, Martinez FJ, Martin N, Singh D, Wise R, Zheng J, Lipson DA. Triple Versus Dual Combination Therapy in Chronic Obstructive Pulmonary Disease in Asian Countries: Analysis of the IMPACT Trial. Pulm Ther. 2021 Jun;7(1):101-118. doi: 10.1007/s41030-020-00136-3. Epub 2020 Nov 17. PMID 33201438
- [Derived] Bourdin A, Criner G, Devouassoux G, Dransfield M, Halpin DMG, Han MK, Jones CE, Kalhan R, Lange P, Lettis S, Lipson DA, Lomas DA, Echave-Sustaeta Maria-Tome JM, Martin N, Martinez FJ, Quasny H, Sail L, Siler TM, Singh D, Thomashow B, Watz H, Wise R, Hanania NA. InforMing the PAthway of COPD Treatment (IMPACT Trial) Single-Inhaler Triple Therapy (Fluticasone Furoate/Umeclidinium/Vilanterol) Versus Fluticasone Furoate/Vilanterol and Umeclidinium/Vilanterol in Patients With COPD: Analysis of the Western Europe and North America Regions. Chronic Obstr Pulm Dis. 2021 Jan;8(1):76-90. doi: 10.15326/jcopdf.2020.0158. PMID 33156982
- [Derived] Zheng J, Zhong N, Wang C, Wei LP, Zhou XD, Zhao L, Dong Yuan Y, He B, Wu B, Du X, Song J, Lipson DA. Single inhaler triple therapy (FF/UMEC/VI) versus FF/VI and UMEC/VI in patients with COPD: subgroup analysis of the China cohort in the IMPACT trial. Curr Med Res Opin. 2021 Jan;37(1):145-155. doi: 10.1080/03007995.2020.1844646. Epub 2020 Dec 7. PMID 33124900
- [Derived] Marin JM, Mateos L, Roldan J, Echave-Sustaeta JM, Pascual-Guardia S, Pardo MV, Velasco B, Jones CE, Kilbride S, Lipson DA. Efficacy of FF/UMEC/VI compared with FF/VI and UMEC/VI in patients with COPD: subgroup analysis of the Spain cohort in IMPACT. Ther Adv Respir Dis. 2020 Jan-Dec;14:1753466620963021. doi: 10.1177/1753466620963021. PMID 33121372
- [Derived] Hanania NA, Mannino DM, Criner GJ, Dransfield MT, Han MK, Jones CE, Kilbride S, Lomas DA, Martin N, Martinez FJ, Singh D, Wise RA, Halpin DMG, Lima R, Lipson DA. Effect of Age on the Efficacy and Safety of Once-Daily Single-Inhaler Triple-Therapy Fluticasone Furoate/Umeclidinium/Vilanterol in Patients With COPD: A Post Hoc Analysis of the Informing the Pathway of COPD Treatment Trial. Chest. 2021 Mar;159(3):985-995. doi: 10.1016/j.chest.2020.09.253. Epub 2020 Oct 5. PMID 33031829
- [Derived] Tabberer M, Jones CE, Kilbride S, Halpin DMG, Lomas DA, Pascoe S, Singh D, Wise RA, Criner GJ, Lange P, Dransfield MT, Han MK, Martinez FJ, Kaisermann MC, Lipson DA. Single-Inhaler Triple Therapy and Health-Related Quality of Life in COPD: The IMPACT Study. Adv Ther. 2020 Sep;37(9):3775-3790. doi: 10.1007/s12325-020-01409-8. Epub 2020 Jul 9. PMID 32647911
- [Derived] Han MK, Criner GJ, Dransfield MT, Halpin DMG, Jones CE, Kilbride S, Lange P, Lettis S, Lipson DA, Lomas DA, Martin N, Wise RA, Singh D, Martinez FJ. The Effect of Inhaled Corticosteroid Withdrawal and Baseline Inhaled Treatment on Exacerbations in the IMPACT Study. A Randomized, Double-Blind, Multicenter Clinical Trial. Am J Respir Crit Care Med. 2020 Nov 1;202(9):1237-1243. doi: 10.1164/rccm.201912-2478OC. PMID 32584168
- [Derived] Day NC, Kumar S, Criner G, Dransfield M, Halpin DMG, Han MK, Jones CE, Kaisermann MC, Kilbride S, Lange P, Lomas DA, Martin N, Martinez FJ, Singh D, Wise R, Lipson DA. Single-inhaler triple therapy fluticasone furoate/umeclidinium/vilanterol versus fluticasone furoate/vilanterol and umeclidinium/vilanterol in patients with COPD: results on cardiovascular safety from the IMPACT trial. Respir Res. 2020 Jun 5;21(1):139. doi: 10.1186/s12931-020-01398-w. PMID 32503599
- [Derived] Bogart MR, Hopson SD, Shih HC, Stanford RH, Coutinho AD. COPD exacerbation costs in the IMPACT study: a within-trial analysis. Am J Manag Care. 2020 May 1;26(5):e150-e154. doi: 10.37765/ajmc.2020.43157. PMID 32436683
- [Derived] Halpin DMG, Dransfield MT, Han MK, Jones CE, Kilbride S, Lange P, Lipson DA, Lomas DA, Martinez FJ, Pascoe S, Singh D, Wise R, Criner GJ. The effect of exacerbation history on outcomes in the IMPACT trial. Eur Respir J. 2020 May 21;55(5):1901921. doi: 10.1183/13993003.01921-2019. Print 2020 May. PMID 32299860
- [Derived] Lipson DA, Crim C, Criner GJ, Day NC, Dransfield MT, Halpin DMG, Han MK, Jones CE, Kilbride S, Lange P, Lomas DA, Lettis S, Manchester P, Martin N, Midwinter D, Morris A, Pascoe SJ, Singh D, Wise RA, Martinez FJ. Reduction in All-Cause Mortality with Fluticasone Furoate/Umeclidinium/Vilanterol in Patients with Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2020 Jun 15;201(12):1508-1516. doi: 10.1164/rccm.201911-2207OC. PMID 32162970
- [Derived] Ismaila AS, Risebrough N, Schroeder M, Shah D, Martin A, Goodall EC, Ndirangu K, Criner G, Dransfield M, Halpin DM, Han MK, Lomas DA. Cost-Effectiveness Of Once-Daily Single-Inhaler Triple Therapy In COPD: The IMPACT Trial. Int J Chron Obstruct Pulmon Dis. 2019 Nov 29;14:2681-2695. doi: 10.2147/COPD.S216072. eCollection 2019. PMID 31819401
- [Derived] Mehta R, Farrell C, Hayes S, Birk R, Okour M, Lipson DA. Population Pharmacokinetic Analysis of Fluticasone Furoate/Umeclidinium Bromide/Vilanterol in Patients with Chronic Obstructive Pulmonary Disease. Clin Pharmacokinet. 2020 Jan;59(1):67-79. doi: 10.1007/s40262-019-00794-w. PMID 31321713
- [Derived] Pascoe S, Barnes N, Brusselle G, Compton C, Criner GJ, Dransfield MT, Halpin DMG, Han MK, Hartley B, Lange P, Lettis S, Lipson DA, Lomas DA, Martinez FJ, Papi A, Roche N, van der Valk RJP, Wise R, Singh D. Blood eosinophils and treatment response with triple and dual combination therapy in chronic obstructive pulmonary disease: analysis of the IMPACT trial. Lancet Respir Med. 2019 Sep;7(9):745-756. doi: 10.1016/S2213-2600(19)30190-0. Epub 2019 Jul 4. PMID 31281061
- [Derived] Lipson DA, Barnhart F, Brealey N, Brooks J, Criner GJ, Day NC, Dransfield MT, Halpin DMG, Han MK, Jones CE, Kilbride S, Lange P, Lomas DA, Martinez FJ, Singh D, Tabberer M, Wise RA, Pascoe SJ; IMPACT Investigators. Once-Daily Single-Inhaler Triple versus Dual Therapy in Patients with COPD. N Engl J Med. 2018 May 3;378(18):1671-1680. doi: 10.1056/NEJMoa1713901. Epub 2018 Apr 18. PMID 29668352
- [Derived] Pascoe SJ, Lipson DA, Locantore N, Barnacle H, Brealey N, Mohindra R, Dransfield MT, Pavord I, Barnes N. A phase III randomised controlled trial of single-dose triple therapy in COPD: the IMPACT protocol. Eur Respir J. 2016 Aug;48(2):320-30. doi: 10.1183/13993003.02165-2015. Epub 2016 Jul 13. PMID 27418551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic obstructive pulmonary disease (COPD), were randomized to the study. Study was conducted from 30 June 2014 to 17 July 2017, at total of 971 sites in 37 countries.
Groups:
- FF/UMEC/VI: The eligible participants in this arm received Fluticasone Furoate (FF)/Umeclidinium (UMEC)/Vilanterol (VI) as a fixed dose combination (FDC) as 100 microgram (µcg)/62.5µcg/25µcg once daily (QD) via a dry powder inhaler (DPI), in the morning, for duration of 52 weeks.
- FF/VI: The eligible participants in this arm received FF/VI 100µcg/25µcg QD via DPI, in the morning for duration of 52 weeks.
- UMEC/VI: The eligible participants in this arm received UMEC/VI 62.5µcg/25µcg QD via DPI, in the morning for duration of 52 weeks.
Period: Overall Study
Arm/Group | FF/UMEC/VI | FF/VI | UMEC/VI
Started | 4151 | 4134 | 2070
Completed Investigational Product (IP) | 3393 | 3094 | 1504
Not Completed IP | 758 | 1040 | 566
Withdrew IP (WIP): Adverse Event | 249 | 325 | 186
WIP: Lack of Efficacy | 163 | 313 | 172
Withdrew IP: Protocol Deviation | 32 | 41 | 19
WIP (Other): Stopping Criteria Reached | 4 | 1 | 2
WIP: Study Closed/Terminated | 5 | 2 | 5
WIP: Lost to Follow-up | 21 | 25 | 14
WIP: Investigator Discretion | 33 | 36 | 15
WIP: Withdrawal by Participant | 250 | 296 | 153
WIP :Did Not Complete Study Treatment | 1 | 1 | 0
Completed | 3714 | 3598 | 1775
Not Completed | 437 | 536 | 295
Not completed — Adverse Event | 162 | 180 | 111
Not completed — Other: Study Closed or terminated | 5 | 2 | 4
Not completed — Lost to Follow-up | 30 | 36 | 22
Not completed — Physician Decision | 47 | 57 | 28
Not completed — Withdrawal by Subject | 192 | 261 | 130
Not completed — Other: Reason not provided by site | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FF/UMEC/VI: The eligible participants in this arm received FF/UMEC/VI as a FDC as 100 µcg/62.5µcg/25µcg, QD via a DPI, in the morning, for duration of 52 weeks.
- Total: Total of all reporting groups
Arm/Group | FF/UMEC/VI | FF/VI | UMEC/VI | Total
Number analyzed (Participants) | 4151 | 4134 | 2070 | 10355
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (8.24) | 65.3 (8.30) | 65.2 (8.26) | 65.3 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1385 | 1386 | 714 | 3485
  Male | 2766 | 2748 | 1356 | 6870
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 87 | 86 | 45 | 218
  Asian - Central/South Asian Heritage | 6 | 3 | 1 | 10
  Asian - East Asian Heritage | 362 | 374 | 177 | 913
  Asian - Japanese Heritage | 151 | 152 | 82 | 385
  Asian - South East Asian Heritage | 149 | 147 | 75 | 371
  Black or African American | 122 | 99 | 43 | 264
  Native Hawaiian or other Pacific Islander | 2 | 3 | 2 | 7
  White - Arabic/North African Heritage | 31 | 45 | 24 | 100
  White - White/Caucasian/European Heritage | 3200 | 3179 | 1604 | 7983
  Multiple | 41 | 45 | 17 | 103
  Unknown | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of On-treatment Moderate/Severe Exacerbations Comparing FF/UMEC/VI With UMEC/VI and FF/VI
Description: The annual rate of moderate or severe COPD exacerbations which occurred during treatment was assessed. Moderate exacerbations were defined as exacerbations that required treatment with oral/systemic corticosteroids and/or antibiotics (not involving hospitalization or resulting in death). Severe exacerbations were defined as exacerbations that required hospitalization or resulted in death. Analysis performed using a generalized linear model assuming a negative binomial distribution. ITT population was used which comprised of all randomized participants, excluding those who were randomized in error. Only those participants with non-missing co-variates were included in the analysis.
Time Frame: Up to Week 52
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per participant per year
Arm/Group | FF/UMEC/VI | FF/VI | UMEC/VI
Number analyzed (Participants) | 4145 | 4133 | 2069
Exacerbations per participant per year | 0.91 [0.87 to 0.95] | 1.07 [1.02 to 1.12] | 1.21 [1.14 to 1.29]
Statistical Analysis 1: Comparison: FF/UMEC/VI vs UMEC/VI; Test type: Superiority; p < 0.001, Negative binomial model — The adjusted p-values should be compared against a reference level of 0.05 in order to infer statistical significance for either of the comparisons; Rate ratio = 0.75, 95% CI 2-sided [0.70 to 0.81] — Covariates of treatment group, sex, exacerbation history (<=1, >=2 moderate/severe), smoking status (Screening), geographical region and post-bronchodilator percent predicted Forced expiratory volume in 1 second (FEV1) (Screening) were used
Statistical Analysis 2: Comparison: FF/UMEC/VI vs FF/VI; Test type: Superiority; p < 0.001, Negative binomial model — [p-value comment as in outcome 1, analysis 1]; Rate ratio = 0.85, 95% CI 2-sided [0.80 to 0.90] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1), at Week 52 Comparing FF/UMEC/VI With FF/VI
Description: FEV1 was defined as the amount of air a person exhales in one second. Change from Baseline was calculated as the value of FEV1 at Week 52 minus the value at Baseline. Baseline for trough FEV1 was defined as Day 1 (Pre-dose). Only those participants with non-missing co-variates were included in the analysis. The analysis was performed using a Repeated measures model with covariates of treatment group, smoking status (Screening), geographical region, visit, Baseline, Baseline by visit and treatment group by visit interactions.
Time Frame: Baseline and Week 52
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | FF/UMEC/VI | FF/VI
Number analyzed (Participants) | 3366 | 3060
Liter | 0.094 (0.0042) | -0.003 (0.0044)
Statistical Analysis 1: Comparison: FF/UMEC/VI vs FF/VI; Test type: Superiority; p < 0.001, Mixed Models Repeated Measures — The adjusted p-value at Week 52 should be compared against a reference level of 0.05 in order to infer statistical significance for the comparison of FF/UMEC/VI versus (vs) FF/VI at Week 52; Mean Difference (Net) = 0.097, 95% CI 2-sided [0.085 to 0.109], Standard Error of Mean 0.0061

3. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire for (SGRQ) Total Score at Week 52 Comparing FF/UMEC/VI With FF/VI
Description: SGRQ is a disease specific-questionnaire, designed to measure impact of respiratory disease and its treatment on a COPD participant's Health Related Quality of Life (HRQoL). SGRQ contains 14 questions with total of 40 items grouped into three domains (Symptoms, Activity, and Impacts). The overall summary score along with scores for the individual domains of symptoms, activity and impacts were assessed. Score was calculated by summing the pre-assigned weights of answers, dividing by sum of maximum weights for items in SGRQ. Total scores ranged from 0 to 100. A decrease in score indicates improvement in HRQoL and higher score implies worse quality of life. Change from Baseline was calculated as total score at Week 52 minus value at Baseline. Baseline was defined as Day 1. Minimum clinically important difference (MCID) for this instrument is a 4-point improvement (decrease from Baseline). Only those participants with non-missing co-variates were included in the analysis.
Time Frame: Baseline and Week 52
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Scores on SGRQ scale
Arm/Group | FF/UMEC/VI | FF/VI
Number analyzed (Participants) | 3318 | 3026
Scores on SGRQ scale | -5.5 (0.23) | -3.7 (0.24)
Statistical Analysis 1: Comparison: FF/UMEC/VI vs FF/VI; Test type: Superiority; p < 0.001, Mixed Models Repeated Measures — The adjusted p-value at Week 52 should be compared against a reference level of 0.05 in order to infer statistical significance for the comparison of FF/UMEC/VI vs FF/VI at Week 52; Mean Difference (Net) = -1.8, 95% CI 2-sided [-2.4 to -1.1], Standard Error of Mean 0.34

4. Secondary Outcome: Time to First On-treatment Moderate/Severe Exacerbation Comparing FF/UMEC/VI With FF/VI and With UMEC/VI
Description: This measures the number of days, to the first onset of moderate or severe exacerbations. Moderate exacerbations, were defined as exacerbations that required treatment with oral/systemic corticosteroids and/or antibiotics (not involving hospitalization or resulting in death). Severe exacerbations, were defined as exacerbations that required hospitalization or resulted in death. The Hazard ratio from Cox proportional hazards model with covariates of treatment group, sex, exacerbation history (<=1, >=2 moderate/severe), smoking status (Screening), geographical region and post-bronchodilator percent predicted FEV1 (Screening), have been reported. Only those participants with non-missing co-variates were included in the analysis. First quartile and median time to onset are taken from the Kaplan-Meier estimates. If <25% (and <50%) of participants experienced the event within a treatment then Q1 (and median) time to onset are displayed as NA (not applicable) for that treatment.
Time Frame: Up to Week 52
Population: ITT Population.
Measure: Number; unit: Days
Arm/Group | FF/UMEC/VI | FF/VI | UMEC/VI
Number analyzed (Participants) | 1959 | 2039 | 1036
Days
  First quartile time to onset | 112 | 81 | 73
  Median time to onset | NA — If <25% (and <50%) of participants experienced the event within a treatment then Q1 (and median) time to onset are displayed as NA (not applicable) for that treatment. | NA — If <25% (and <50%) of participants experienced the event within a treatment then Q1 (and median) time to onset are displayed as NA (not applicable) for that treatment. | 306
Statistical Analysis 1: Comparison: FF/UMEC/VI vs FF/VI; Test type: Superiority; p < 0.001, Cox proportional hazard model — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.80 to 0.91]
Statistical Analysis 2: Comparison: FF/UMEC/VI vs UMEC/VI; Test type: Superiority; p < 0.001, Cox proportional hazard model; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.78 to 0.91]

5. Secondary Outcome: Annual Rate of On-treatment Moderate/Severe Exacerbations Comparing FF/UMEC/VI With UMEC/VI in the Subset of Participants With a Blood Eosinophil Count >=150 Cells Per Microliter
Description: The annual rate of moderate or severe COPD exacerbations during the treatment, for participants with blood eosinophil count >=150 cells per microliter , has been reported. Moderate exacerbations, were defined as exacerbations that required treatment with oral/systemic corticosteroids and/or antibiotics (not involving hospitalization or resulting in death). Severe exacerbations were defined as exacerbations that required hospitalization or resulted in death. Only those participants with non-missing co-variates and non-missing eosinophil, at Baseline were included in the analysis.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per participant per year
Arm/Group | FF/UMEC/VI | UMEC/VI
Number analyzed (Participants) | 2296 | 1195
Exacerbations per participant per year | 0.95 [0.90 to 1.01] | 1.39 [1.29 to 1.51]
Statistical Analysis 1: Comparison: FF/UMEC/VI vs UMEC/VI; Test type: Superiority; p < 0.001, Negative binomial Model; Rate ratio = 0.68, 95% CI 2-sided [0.62 to 0.75]

6. Secondary Outcome: Time to First On-treatment Moderate/Severe Exacerbation Comparing FF/UMEC/VI With UMEC/VI in the Subset of Particpants With a Blood Eosinophil Count >=150 Cells Per Microliter at Baseline
Description: This measures the number of days, to the first onset of moderate or severe exacerbations for participants with blood eosinophil count >=150 cells per microliter, at Baseline has been reported. Moderate exacerbations, were defined as exacerbations that required treatment with oral/systemic corticosteroids and/or antibiotics (not involving hospitalization or resulting in death). Severe exacerbations, were defined as exacerbations that required hospitalization or resulted in death. Only those participants with non-missing co-variates and non missing eosinophils at Baseline were included in the analysis. First quartile and median time to onset are taken from the Kaplan-Meier estimates. If <25% (and <50%) of participants experienced the event within a treatment then Q1 (and median) time to onset are displayed as NA (not applicable) for that treatment.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Days
Arm/Group | FF/UMEC/VI | UMEC/VI
Number analyzed (Participants) | 2296 | 1195
Days
  First quartile time to onset | 107 | 55
  Median time to onset | NA — If <25% (and <50%) of participants experienced the event within a treatment then Q1 (and median) time to onset are displayed as NA (not applicable) for that treatment. | 253
Statistical Analysis 1: Comparison: FF/UMEC/VI vs UMEC/VI; Test type: Superiority; p < 0.001, Cox proportional hazard model; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.70 to 0.85]

7. Secondary Outcome: Annual Rate of On-treatment Severe Exacerbations Comparing FF/UMEC/VI With FF/VI and With UMEC/VI
Description: The annual rate of severe COPD exacerbations during the treatment, has been reported. Severe exacerbations were defined as exacerbations that required hospitalization or resulted in death. The covariates of treatment group, sex, exacerbation history (<=1, >=2 moderate/severe), smoking status (Screening), geographical region and post-bronchodilator percent predicted FEV1 (Screening) were used. Only those participants with non-missing co-variates were included in the analysis
Time Frame: Up to Week 52
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per participant per year
Arm/Group | FF/UMEC/VI | FF/VI | UMEC/VI
Number analyzed (Participants) | 4145 | 4133 | 2069
Exacerbations per participant per year | 0.13 [0.12 to 0.14] | 0.15 [0.13 to 0.16] | 0.19 [0.17 to 0.22]
Statistical Analysis 1: Comparison: FF/UMEC/VI vs FF/VI; Test type: Superiority; p = 0.064, Negative binomial model; Rate Ratio = 0.87, 95% CI 2-sided [0.76 to 1.01]
Statistical Analysis 2: Comparison: FF/UMEC/VI vs UMEC/VI; Test type: Superiority; p < 0.001, Negative binomial model; Rate ratio = 0.66, 95% CI 2-sided [0.56 to 0.78]

ADVERSE EVENTS:
Time Frame: On-treatment Serious adverse events (SAEs) and Adverse events (AEs) are reported from the first dose of randomized medication up to Week 52.
Description: All AEs and SAEs in the ITT Population were reported. The number of on-treatment deaths are reported from date of first dose of study medication up to the day after the last date of study medication.
Groups:
- FF/UMEC/VI 100/62.5/25: The eligible participants in this arm received FF/UMEC/VI as a FDC as 100 µcg/62.5µcg/25µcg, QD via a DPI, in the morning, for duration of 52 weeks.
- FF/VI 100/25: The eligible participants in this arm received FF/VI 100µcg/25µcg QD via DPI, in the morning for duration of 52 weeks.
- UMEC/VI 62.5/25: The eligible participants in this arm received UMEC/VI 62.5µcg/25µcg QD via DPI, in the morning for duration of 52 weeks.
Arm/Group | FF/UMEC/VI 100/62.5/25 | FF/VI 100/25 | UMEC/VI 62.5/25
All-Cause Mortality (participants affected / at risk) | 68/4151 | 76/4134 | 49/2070
Serious Adverse Events (participants affected / at risk) | 895/4151 | 850/4134 | 470/2070
Other Adverse Events (participants affected / at risk) | 1389/4151 | 1278/4134 | 596/2070
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF/UMEC/VI 100/62.5/25 (N=4151) | FF/VI 100/25 (N=4134) | UMEC/VI 62.5/25 (N=2070)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 3 (3) | 3 (3)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 13 (14) | 8 (8) | 6 (6)
Angina pectoris (Cardiac disorders) | 2 (3) | 3 (3) | 2 (2)
Angina unstable (Cardiac disorders) | 7 (8) | 6 (6) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 21 (24) | 13 (13) | 6 (6)
Atrial flutter (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Atrioventricular dissociation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (4) | 2 (2) | 2 (2)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 12 (12) | 7 (8) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 2 (3) | 2 (2) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 21 (28) | 12 (12) | 7 (10)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 4 (4) | 4 (4) | 5 (5)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cor pulmonale chronic (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 4 (4) | 2 (2) | 3 (3)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 10 (10) | 6 (6) | 7 (7)
Myocardial ischaemia (Cardiac disorders) | 5 (6) | 1 (1) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial bridging (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Odontogenic cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Amaurosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 3 (3) | 5 (5) | 2 (2)
Cataract nuclear (Eye disorders) | 2 (3) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (3) | 3 (3) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 4 (5) | 2 (2) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 6 (6) | 4 (4) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Retroperitoneal fibrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 5 (5) | 3 (3) | 7 (7)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 3 (3) | 5 (5) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site fibrosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Medical device site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 8 (8) | 10 (10) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 2 (2)
Stent-graft endoleak (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 2 (2)
Sudden death (General disorders) | 3 (3) | 2 (2) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 3 (3) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 5 (5)
Gallbladder perforation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 2 (2)
Anaphylactic shock (Immune system disorders) | 2 (2) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 10 (10) | 10 (11) | 3 (3)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 6 (6) | 1 (4) | 3 (3)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
Empyema (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 5 (5) | 2 (2)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haemophilus infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected varicose vein (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 8 (8) | 19 (20) | 7 (8)
Influenza (Infections and infestations) | 7 (7) | 6 (6) | 5 (5)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 7 (8) | 4 (4) | 4 (5)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mycoplasma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nosocomial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 184 (198) | 152 (165) | 54 (55)
Pneumonia bacterial (Infections and infestations) | 2 (3) | 9 (9) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 9 (10) | 8 (8) | 6 (6)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 4 (4) | 2 (2) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subacute endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 7 (7) | 4 (4)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Conjunctival laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 9 (10) | 3 (3) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Biopsy prostate (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Streptococcus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Acetonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 2 (2)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 0 (0)
Bone infarction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 3 (3)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (4) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 5 (6) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign fallopian tube neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (5) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Bladder transitional cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 2 (2)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1)
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Epiglottic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0)
Haemangioma of spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hepatic angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 0 (0)
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 10 (10) | 2 (2)
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain stem ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral amyloid angiopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 7 (7) | 6 (7) | 3 (3)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 4 (4) | 5 (5) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mental impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral nerve paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Radicular syndrome (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Simple partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 6 (6) | 5 (5) | 3 (3)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 8 (8) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (3)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 4 (4) | 1 (1)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 9 (9) | 6 (9)
Bladder disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 3 (3) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 3 (4) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal aneurysm (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal cyst haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 3 (4) | 2 (2)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (3) | 1 (1) | 2 (2)
Vesicocutaneous fistula (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 2 (2)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 23 (27) | 17 (17) | 16 (20)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 443 (554) | 450 (569) | 269 (337)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 11 (12) | 3 (3)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (5) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7) | 6 (6)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 22 (23) | 21 (21) | 7 (7)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Peau d'orange (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Acute aortic syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 3 (3) | 1 (1)
Embolism arterial (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 2 (3) | 2 (2)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 2 (2) | 2 (2)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Varicose ulceration (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF/UMEC/VI 100/62.5/25 (N=4151) | FF/VI 100/25 (N=4134) | UMEC/VI 62.5/25 (N=2070)
Viral upper respiratory tract infection (Infections and infestations) | 520 (712) | 479 (658) | 222 (316)
Upper respiratory tract infection (Infections and infestations) | 297 (401) | 283 (383) | 117 (162)
Oral candidiasis (Infections and infestations) | 161 (203) | 146 (176) | 41 (50)
Bronchitis (Infections and infestations) | 142 (165) | 120 (152) | 70 (83)
Pneumonia (Infections and infestations) | 121 (131) | 127 (135) | 41 (43)
Headache (Nervous system disorders) | 233 (385) | 197 (332) | 101 (139)
Back pain (Musculoskeletal and connective tissue disorders) | 146 (180) | 139 (164) | 83 (101)
Cough (Respiratory, thoracic and mediastinal disorders) | 145 (168) | 117 (128) | 58 (75)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT02164513/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT02164513/SAP_001.pdf